CLINICAL TRIAL: NCT01322906
Title: Allogeneic Bone Marrow Mesenchymal Stem Cells Transplantation in Patients With Liver Failure Caused by HBV
Brief Title: Allogeneic Bone Marrow Mesenchymal Stem Cells Transplantation in Patients With Liver Failure Caused by Hepatitis B Virus (HBV)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Lin Bingliang, Third Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABMS-LF
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2010-10

CONDITIONS: Liver Failure
Keywords: ABMLF; Allogenic Bone marrow Mesenchymal Stem Cells; Liver Failure; Transplantation
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group A (Other): Thirty of the enrolled patients were assigned to Group A to receive comprehensive treatment including antiviral drugs, lowering aminotransferase and jaundice medicine.
  Interventions: Other: Group 1; Other: Group 2; Other: Group 3

INTERVENTIONS:
Other: Group 1 — Thirty of the enrolled patients were assigned to Group B to receive comprehensive treatment, as well as allogeneic bone marrow mesenchymal stem cells transplantation by peripheral vein(2×105/Kg, once a week, 4 times).
Other: Group 2 — Thirty of the enrolled patients were assigned to Group B to receive comprehensive treatment, as well as allogeneic bone marrow mesenchymal stem cells transplantation by peripheral vein(1×106/Kg, once a week, 4 times).
Other: Group 3 — Thirty of the enrolled patients were assigned to Group B to receive comprehensive treatment, as well as allogeneic bone marrow mesenchymal stem cells transplantation by peripheral vein(5×106/Kg, once a week, 4 times).

SUMMARY:
Allogeneic Bone Marrow Mesenchymal Stem Cells Transplantation in Patients with Liver Failure Caused by hepatitis B virus (HBV)

ELIGIBILITY:
Inclusion Criteria:

* Liver failure caused by HBV
* Model for End-Stage Liver Disease (MELD) < 30

Exclusion Criteria:

* Liver Failure caused by other reasons, such as autoimmune diseases, alcohol, drug and so on.
* History of moderate to severe hepatic encephalopathy or variceal bleeding during the last two months before enrollment.
* Severe problems in other vital organs (e.g.the heart,renal or lungs).
* Tumor on ultrasonography, CT or MRI examination.
* Pregnant or lactating women.
* HIV infection.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-11 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Liver Function | 12months
  The levels of serum alanine aminotransferase (ALT), aspartate aminotransferase(AST),total bilirubin (TB),prothrombin time (PT), prothrombin activity(PTA),INR,albumin (ALB),globulin(GLB), prealbumin(PA),creatinine(Cr), Urea nitrogen(BUN),number of leucocyte,erythrocyte and platelet, cytokines,liver histological
Immune state | 12months
  cytokine